CLINICAL TRIAL: NCT05685446
Title: Gastric Emptying and Gastric Volume After Ingestion of 175 ml of Ice Water Prior to Elective Gastroscopy in Healthy Adults
Brief Title: Gastric Volume After Drinking 175 ml of Ice Water Prior to Gastroscopy in Healthy Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Caroline Hornnes Pedersen, MD, Regionshospital Nordjylland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20190056
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Fasting; Perioperative Pulmonary Aspiration
Keywords: Gastroscopy; Gastric volume; Anaesthesia
MeSH Terms: conditions — Fasting | interventions — major intrinsic protein, plant

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 175 ml ice water (Experimental): Ingestion of 175 ml ice water 15 minutes prior to gastroscopy
  Interventions: Other: Ice water
- Fasting (No Intervention): Continued fasting

INTERVENTIONS:
Other: Ice water — Ingestion of 175 ml iced tap water 15 minutes prior to elective gastroscopy
  Other Names: Iced tap water
  Arms: 175 ml ice water

SUMMARY:
Recommendation for fluid fasting is two hours prior to anaesthesia, however, less may be acceptable. The current study compares ingestion of 175 ml ice water prior to elective gastroscopy vs. standard fasting on gastric residual volume.

DETAILED DESCRIPTION:
Recommendations regarding fasting requirements prior to general anaesthesia is two hours for fluids. Recent research indicates that reduced fluid fasting time may be acceptable. The current study aimed to compare ingestion of 175 ml ice water 15 minutes prior to procedure compared to standardized fasting regimen on residual gastric volumes in patients receiving elective gastroscopy, as these volumes may have implications for fasting requirements.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective gastroscopy in a medical outpatient clinic
* American Society of Anesthesiologists physical status classification system category (ASA score) I or II
* Age 18 years or above

Exclusion Criteria:

* Any increased risk of aspiration, eg. dysphagia, previous aspiration, non-fasting status, or known alcohol abuse
* Suspected delayed gastric emptying, eg. regular opioid use within three days
* Enteral pre-medication required
* Any structural gastric or esophageal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume | 15 minutes
  Aspired residual gastric fluid volume at start of gastroscopy

SECONDARY OUTCOMES:
Nausea and dyspepsia | 15 minutes
  Proportion of patients reporting nausea or dyspeptic symptoms prior to gastroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Damgaard, MD, PhD, Study Chair — Regional Hospital of Northern Denmark, Hjørring
Locations (1):
- Department of Anaestesia, Hjørring, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No